CLINICAL TRIAL: NCT01272154
Title: Cerebellum and Cortical Plasticity: the Case of Dystonia
Acronym: CERDYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Sree Chitra Tirunal Institute for Medical Sciences & Technology (Other Government); Policlinico G . Martino, Messina Italy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: C10-01; 2010-A00931-38 (Registry Identifier: IDRCB)
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-01

CONDITIONS: Dystonia
Keywords: Cerebellum; Cortical plasticity; Sensorimotor adaptation; Dystonia; Cerebral Palsy; Transcranial Magnetic Stimulation; and
MeSH Terms: conditions — Dystonia; Cerebral Palsy | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Primary cervical dystonia Patients (Experimental)
  Interventions: Other: Transcranial magnetic stimulation
- Primary upperlimb Dystonia Patients (Experimental)
  Interventions: Other: Transcranial magnetic stimulation
- Secondary Cervical or Upperlimb Dystonia due to cerebral palsy (Experimental)
  Interventions: Other: Transcranial magnetic stimulation
- Healthy volunteers (Other)
  Interventions: Other: Transcranial magnetic stimulation

INTERVENTIONS:
Other: Transcranial magnetic stimulation — Transcranial magnetic stimulation (PAS and rTMS)

SUMMARY:
Purpose

- Objective : Sensorimotor adaptation allows the modification of the motor command taking into account the errors detected during execution of prior movements. It involves a large cortico-subcortical network. Isolated lesions of this network do not systematically alter sensorimotor adaptation except for cerebellar lesions. The cerebellum is thus a key structure for sensorimotor adaptation. However, the link between cerebellar and the cortical plasticity underlying sensorimotor adaptation remain unknown. Alteration of sensorimotor adaptation is associated with dystonia but it is unclear whether it is a cause or consequence of dystonia. It has been hypothesized that the abnormal plasticity observed in dystonia could account for the associated alteration of sensorimotor adaptation.

Classically, basal ganglia dysfunction is considered to be crucial for dystonia pathogenesis. However, recent studies suggest that the involvement of the cerebellum may also be important in this setting. In primary dystonia, imaging studies showed abnormal cerebellar activation during sensorimotor adaptation tasks and neurophysiological studies demonstrated a decrease of cerebellar output.

The aim of this study is to investigate the role of the cerebellum in the cortical plasticity underlying sensorimotor adaptation both in healthy subjects (normal plasticity) and in dystonic patients (abnormal plasticity).

- Methods: Paired associative stimulation PAS consists in repetitive pairing of a peripheral nerve and a cortical stimulation. This kind of stimulation has been designed to induce artificial plasticity that can be easily measured. This PAS induced sensorimotor plasticity is exacerbated and has lost its topographical specificity in dystonic patients.TMS using trains of TMS pulses (rTMS) can be applied on the cerebellum to modulate its output. We will test the effect of rTMS induced modulation (cTBS- inhibitory, iTBS-excitatory, sham) of the cerebellar output on PAS induced plasticity in patients with dystonia and healthy control.

We will also assess the acute effect of the rTMS induced modulation of the cerebellar output on the dystonic symptoms and on the performance at a validated sensorimotor adaptation task. This will be done by double blind post-hoc scoring of the dystonia (BFM or TWSTRS) on standardized videorecording and measurement of the performance at the task after each rTMS session (cTBS, iTBS, sham).

Finally, we will assess the variation of PAS effect on other parameters reflecting cortical excitability after each rTMS session (cTBS, iTBS, sham).

ELIGIBILITY:
Inclusion criteria

All subjects

* Age >18 years and < 70 years
* Normal physical and neurological examination, except for dystonia (when present)
* No treatment with botulinum toxin during the last three months
* No treatment altering the cortical excitability
* Agreement to use a medically acceptable method of contraception throughout the study for female of childbearing potential

Primary focal dystonia group

* Patients with cervical and/or upper limb dystonia
* No cause of secondary dystonia

Secondary dystonia group

• Cervical dystonia and/or upper limb dystonia History of perinatal anoxia

Exclusion criteria

* MMS ≤ 24/30
* Current neurological or psychiatric illness other than dystonia.
* Individual who is on medication which is known to lower seizure threshold (see lists above), or who has a pacemaker, an implanted medical pump, a metal plate, a metal plate or metal object in the skull or eye (for example after brain surgery) will be excluded
* Uncontrollable medical problems not related to dystonia such as; cardiopulmonary disease, severe rheumatoid arthritis, active joint deformity of arthritic origin, active cancer, or renal disease
* Previous history of seizure(s) or current active epilepsy
* Pregnancy, breast feeding women and women who are of childbearing age and not practicing adequate birth control.
* Patients legally protected
* Patients who are not enrolled at social security

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2012-10-24 (Actual); Study Completion 2012-10-24 (Actual)

PRIMARY OUTCOMES:
Comparison of MEP0/MEP10 and MEP0/MEP30 values obtained after sham, cRTBS or iTBS of the cerebellum. | 6 weeks
  The effect of rTMS induced modulation of the cerebellar output on the PAS induced plasticity will be assessed by measurement of the size variation of a 1mV test motor evoked potential (which reflect cortical excitability) before (MEP0) and 10 and 30 minutes (MEP10 and MEP30) after PAS. The primary outcome measure will be the comparison of MEP0/MEP10 and MEP0/MEP30 values obtained after sham, cRTBS or iTBS of the cerebellum.

SECONDARY OUTCOMES:
Variation of the appropriate dystonic clinical score (depending on the type of dystonia) after each rTMS session (cTBS, iTBS, sham). | 6 weeks
  The effect of rTMS induced modulation of the cerebellar output on dystonic symptoms will be assessed by the variation of the appropriate dystonic clinical score (depending on the type of dystonia) after each rTMS session (cTBS, iTBS, sham).
Measurement of number of errors, mean time to reach the target after each rTMS session (cTBS, iTBS, sham). | 6 weeks
  The effect of rTMS induced modulation of the cerebellar output on the performance at the sensorimotor adaptation task will be assessed by measurement of number of errors, mean time to reach the target after each rTMS session (cTBS, iTBS, sham).
Measurement of the variation of the motor threshold, intracortical inhibition and intracortical facilitation after each rTMS session (cTBS, iTBS, sham). | 6 weeks
  The effect of rTMS induced modulation of the cerebellar output on other parameter reflecting cortical excitability will be assessed by measurement of the variation of the motor threshold, intracortical inhibition and intracortical facilitation after each rTMS session (cTBS, iTBS, sham).

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Roze, MD, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France; Asha Kishore, MD, Principal Investigator — Sree Chitra Tirunal Institute for Medical Sciences and Technology (SCTIMST); Margherita Russo, MD, Principal Investigator — Policlinico G . Martino
Locations (1):
- Hpôpital Pitié Sapétrière - U 975 Plate forme " Pole Exploration de l'homme : Gait, Equilibrium, Posture, and Movement ", Paris, France

REFERENCES:
- [Background] Hubsch C, Roze E, Popa T, Russo M, Balachandran A, Pradeep S, Mueller F, Brochard V, Quartarone A, Degos B, Vidailhet M, Kishore A, Meunier S. Defective cerebellar control of cortical plasticity in writer's cramp. Brain. 2013 Jul;136(Pt 7):2050-62. doi: 10.1093/brain/awt147. PMID 23801734